CLINICAL TRIAL: NCT01100047
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD5069 in Healthy Japanese Subjects After Single and Multiple Ascending Doses
Brief Title: Japanese Single and Multiple Ascending Dose (JSMAD), Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) Study of AZD5069
Acronym: JSMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3550C00005; 2009-018185-35 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-04-08 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Phase I; Japanese healthy volunteer; AZD5069
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD5069
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5069 — Oral suspension
  Arms: 1
Drug: Placebo — Oral suspension
  Arms: 2

SUMMARY:
This is a study in Japanese healthy volunteers to determine the safety and tolerability of the compound, AZD5069. It will also assess how the body handles the drug and how it responds to the drug following single and multiple doses up to 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects with suitable veins for cannulation or repeated venepuncture.
* Have a body mass index (BMI) between 17 and 27 kg/m2 and a body weight between 45 and 80 kg
* Male subjects should be willing to use barrier contraception ie, condoms with spermicide, from the first day of dosing until 3 months after the last dose of investigational product

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness/infection or medical/surgical procedure or trauma, as judged by the Principal Investigator, within 4 weeks of the first administration of investigational product.
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the Investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Adverse events, electrocardiograms (ECGs), laboratory variables, blood pressure, pulse rate, body temperature, QT interval and continuous cardiac monitoring using telemetry | From screening period to follow-up visit 42 days (Maximum)

SECONDARY OUTCOMES:
Assessment of ex vivo GROa stimulated CD11b expression on neutrophils in whole blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose
Measurement of the effect of AZD5069 on blood cells | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose
Pharmacokinetic profile: concentration of AZD5069 in blood | Baselines at Visit 1 or pre-dose Day 1, assessments Visit 2, post-dose until 96hr post final dose. Follow up assessments at Visit 3. Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, Lorch, MD MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Research Site, Croydon, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1336&filename=D3550C00005_Study_Synopsis.pdf